CLINICAL TRIAL: NCT04396262
Title: Effect of Hydro-Thermodynamic (HTD) Processed Blueberries on Postprandial Blood Glucose Control and Antioxidant Status in Human Adults
Brief Title: Effect of Processed Blueberry on Blood Glucose and Antioxidant Status in Human Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-204; 2015-102 (Other: Mount Saint Vincent University)
Record Dates: First submitted 2020-04-01; First posted 2020-05-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Blood Glucose
Keywords: Blueberry; Blood Glucose; Antioxidants; Hydro-Thermodynamic Processing; Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTD-blueberry beverage with white bread (Experimental): The beverage prepared using hydro-thermodynamic processing of whole wild blueberries.
  Interventions: Other: Food-1
- Sweetened water (control) with white bread (Experimental): The water control of the same volume and with the same amount of available carbohydrate as HTD-blueberry beverage.
  Interventions: Other: Food-2

INTERVENTIONS:
Other: Food-1 — HTD-blueberry beverage with white bread.
  Arms: HTD-blueberry beverage with white bread
Other: Food-2 — Sweetened water with white bread as a control.
  Arms: Sweetened water (control) with white bread

SUMMARY:
Canada's Food Guide (2007) recommended 7-10 servings of fruits and vegetables per day for a normal adult population. Although fruit juice (125 ml) is considered as one serving of fruits, the consumption of some fruit juices may be limited due to their high amount of sugar. The consumption of sugary drinks can lead to a rapid rise in postprandial glycaemia. Wild blueberries, due to their high level of anthocyanins, may provide multiple health benefits including improved blood glucose control, however, the consumption of fresh berries is limited by their short seasonal availability. Hydro-Thermodynamic (HTD) processing of blueberries allows the processing of whole berries including their skin and seeds into a beverage with the amount of anthocyanins comparable with fresh berries. The objective of the study is to investigate the effect of HTD-processed blueberries on postprandial glycaemia and antioxidant activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Body mass index (BMI) within normal range (18.5-24.9 kg/m2 for adults)

Exclusion Criteria:

* Chronic metabolic diseases or inflammatory conditions
* Smokers
* A medication that influences glucose control or gastrointestinal function
* Known allergies
* Intellectual disabilities

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 0-120 min
  The concentration of glucose in venous blood after consuming HTD-blueberry beverage with white bread or water control with white bread.

SECONDARY OUTCOMES:
Postprandial antioxidant activity in blood | 0-120 min
  The total antioxidant activity in blood plasma determined using a commercial Antioxidant Assay Kit.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No